CLINICAL TRIAL: NCT03980808
Title: American Sign Language-Accessible Diabetes Education
Acronym: ASL-ADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: H19229; 5P30DK111024-04 (NIH)
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2022-08

CONDITIONS: Diabetes; Deafness
Keywords: Diabetes; Deafness
MeSH Terms: conditions — Diabetes Mellitus; Deafness

STUDY DESIGN:
Intervention Model Description: Quasi-experimental pre and post-test design. There will be one intervention group and one control group as detailed below:
  The intervention group will take the pretest, view the video intervention, take the posttest, and at 30-days following take another posttest.
  The control group will take the pretest and posttest, and at 30-days following take another posttest.
  For those that are assigned to the control groups, at the completion of the study they will be offered the opportunity to view the ASL-ADE intervention.
  The study model was revised to not use the Solomon-Four Group Design because the initial decision to use that design was to measure if there was a pre-test effect. There were no effects for the pre and post-test measures; therefore, we combined the arms into an intervention/no-intervention group, aligning with the primary outcome measures: (1) health literacy, and (2) related health behaviors. The original submission indicated a two-arm study, not a four-arm.
Who Masked: Participant
Masking Description: Participants will not know until the conclusion of the study if they were in the intervention group or the control group. Those on the control group will be offered the opportunity to view the video intervention when data collection concludes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASL-ADE Intervention Arm (Experimental): One-half of enrolled participants will view the ASL-ADE video intervention.
  Interventions: Behavioral: American Sign Language-Accessible Diabetes Education
- Control Arm (Sham Comparator): One-half of enrolled participants will view a non-health related video approximately the same length as the video intervention.
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: American Sign Language-Accessible Diabetes Education — Video-based ASL interpreted diabetes educational intervention (ASL-ADE), the content of which will be derived from diabetes health information regarding symptoms and risk factors that are published by the U.S. Centers for Diseases Control and Prevention (CDC) and the National Institute for Health (NIH) National Diabetes Education Program.
  Other Names: ASL-ADE
  Arms: ASL-ADE Intervention Arm
Behavioral: Control Intervention — Non-health related video approximately the same length as ASL-ADE.
  Arms: Control Arm

SUMMARY:
ASL-ADE will evaluate the efficacy of an ASL-interpreted diabetes educational intervention to the end of improving the health literacy of the target population and addressing their disparate health outcomes.

DETAILED DESCRIPTION:
Georgia Tech's Center for Advanced Communications Policy (CACP) proposes the American Sign Language Accessible Diabetes Education (ASL-ADE) project in response to the Georgia Center for Diabetes Translation Research for a pilot and feasibility study on "Type II translation research in diabetes care and prevention." ASL-ADE will conduct an efficacy study, in the Engagement and Behavior Change Core, with the long-term objective of improved health outcomes for individuals who are Deaf and primarily communicate using ASL. The project will demonstrate the need for diabetes educational materials to be accessible to people who are Deaf and rely on ASL for clear and effective communications. ASL is a distinct language used by individuals of the Deaf community and is grammatically dissimilar to English. Some people who are Deaf rely primarily on ASL and have limited English proficiency. , Other people who are deaf are comfortable with written English. Due to the language diversity within this community, diabetes health education materials are not always accessible. For example, there are low levels of general health literacy among people who are Deaf which increases risk for developing chronic illnesses, , , including diabetes. As such, people who are Deaf also have an increased risk for acute complications associated with diabetes. The low level of health literacy among the target population is directly related to communication/language barriers, as much of the health education outreach mechanisms are exclusionary because of their use of audio and print materials. The hearing population can benefit from incidental learning such as overhearing conversations and watching the news, even commercials. It is a form of socialization that is often taken for granted by people who can hear. To address this access gap, the goals of ASL-ADE are to provide accessible materials to improve health literacy and (1) impact awareness of risk factors, preventive measures, and diabetes symptoms, and (2) elicit the desired behavioral response to seek medical care and modify health-related behaviors. The proposed project will produce a video-based ASL interpreted diabetes educational intervention, and using a pretest-posttest (immediate) 30-day posttest quasi-experimental design, evaluate the effect of the educational intervention on knowledge about diabetes and related health behavior changes. Data will be analyzed along the dimensions of diagnosis status to measure if there is variance in scores for people who are Deaf with a diabetes diagnosis compared to their non-diagnosed counterparts; the a priori hypothesis being that given the communication barriers experienced by people who are Deaf, that no significant between-group differences will be found on pretest scores based on diagnosis status.

This description is revised to exclude analysis along the dimensions of age because our sample did not contain enough subjects between the ages of 18-30 to run a comparison.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Deaf
* Primary language is American Sign Language
* Approximately one-half of the sample must have a diabetes diagnosis.

Exclusion Criteria:

* Minors
* People whose primary language is not ASL
* Individuals unable to provide consent due to impaired decision-making

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muslimah "Salimah" S LaForce, Principal Investigator — Georgia Institute of Technology
Locations (2):
- United States (2):
  - Center for Advanced Communications Policy, Atlanta, Georgia
  - Deaf Link, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data will be submitted to the Inter-university Consortium for Political and Social Research (ICPSR) to allow open, equitable and effective use of the data. Within the ICPSR, we anticipate our data will closely align with existing collections related to Behavioral Sciences, Health Management and Policy, and Disability Concerns. Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared. Other documents to be shared include the study protocol and statistical analysis. These items will be shared immediately following publication (and with no end date) with researchers who provide a methodologically sound proposal for the purpose of achieving the aims of the proposal. Proposals should be directed to salimah@cacp.gatech.edu. To gain access, data requestors will need to sign a data access agreement. Data are available at a third-party website.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available immediately following publication and with no end date.
Access Criteria: The data and supporting information will be shared with researchers who provide a methodologically sound proposal for the purpose of achieving the aims of the proposal. Proposals should be directed to salimah@cacp.gatech.edu. To gain access, data requestors will need to sign a data access agreement. Data are available at a third-party website (Link to be included).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment began on October 27, 2020. Participants were recruited from DeafLink's nationwide reach into the Deaf community.
Period: Overall Study
Arm/Group | ASL-ADE Intervention Arm | Control Arm
Started | 24 | 17
Phase 2 - 30-day Follow-up | 24 | 17
Completed | 22 | 15
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: Adults who are Deaf and whose primary language is Americal Sign Language (ASL), some with a diabetes diagnosis and some without. Participants were randomly assigned to either an intervention group or a control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | ASL-ADE Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 24 | 17 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 15 | 35
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.42 (12.33) | 50.47 (12.76) | 51.6 (12.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 14 | 12 | 26
  Non-Binary | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Indian | 5 | 2 | 7
  Black, African American, or West Indian | 3 | 2 | 5
  Hispanic, Latino or Spanish Origin, regardless of race | 5 | 4 | 9
  More than one race | 4 | 5 | 9
  White or Caucasian | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 24 | 17 | 41
Deaf [Count of Participants; unit: Participants] | 24 | 17 | 41
Diabetes Diagnosis (Yes) [Count of Participants; unit: Participants] | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Health Literacy Score
Description: Data were collected using a study-specific, knowledge-based Diabetes Health Literacy measure which included 15 forced-choice, closed-ended questions to allow for a total score ranging from 0 to 15, with higher scores reflecting better diabetes health literacy. Analysis of change of knowledge compared differences between the intervention arm and the control arm as measured by the changes to the composite scores of the knowledge-based test. One factor Analysis of Variance (ANOVA) was used to calculate the differences with an a priori alpha level of 0.05.
Time Frame: The outcome measure results reflect a comparison of the pre and posttest immediate scores.
Population: Group 1 and Group 2 consisted of adults with and without diabetes who primarily use American Sign Language (ASL) for Communication
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ASL-ADE Intervention Arm | Control Arm
Number analyzed (Participants) | 24 | 17
score on a scale | 1.30 [-.05 to 2.65] | 1.38 [-1.15 to 3.90]
Statistical Analysis 1: Comparison: ASL-ADE Intervention Arm vs Control Arm; Composite scores were calculated for the knowledge based tests. Differences in the pre and post test composite scores were compared using ANOVA. We tested the null hypothesis that score changes in the intervention group and control group were the same; Test type: Equivalence — A priori significance levels were set to 0.05. As this was a pilot study on a demonstration intervention, power analysis were not performed; p = 0.95, ANOVA; Total degrees of freedom (dof) = 17, with between groups dof = 1 and within groups dof = 16; Mean Difference (Net) = 1.33, Standard Error of Mean 0.560

2. Primary Outcome: Frequency of Engagement in Diabetes-Related Health Behaviors
Description: Data were collected using a study-specific questionnaire titled Your Health Behaviors that measure the frequency of diabetes-related health behaviors for a total score ranging from 7 to 35. Each of the diabetes behaviors (physical activity, work physical activity, cigarettes, smoking cessation, alcohol consumption, vegetable consumption, fruit consumption, grain consumption, junk food consumption, fast food consumption) had multiple choice answers that were scaled from 1 - n, with n being the number of options. The least healthy choice was assigned "1", the most healthy choice was assigned "n". Analysis of change in behavior compared differences between the intervention arm and the control arm as measured by the changes in the composite scores of the behavioral intervention. One factor Analysis of Variance (ANOVA) was used to compare the differences with an a priori level of 0.05.
Time Frame: The outcome measure results for the Your Health Behaviors measure are a comparison between the pretest and the 30-day follow-up.
Population: The population consists of people with and without Diabetes who were Deaf who rely on ASL for communication.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ASL-ADE Intervention Arm | Control Arm
Number analyzed (Participants) | 24 | 17
score on a scale | .2381 [-1.1343 to 2.6205] | 2.0625 [0.2532 to 3.8718]
Statistical Analysis 1: Comparison: ASL-ADE Intervention Arm vs Control Arm; Composite scores were calculated for the behavioral self-report tests tests. Differences in the pre and post test composite scores were compared using ANOVA. We tested the null hypothesis that score changes in the intervention group and control group were the same; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.093, ANOVA; Mean Difference (Net) = 1.03, Standard Error of Mean 0.53760

ADVERSE EVENTS:
Time Frame: 3 months.
Arm/Group | ASL-ADE Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/17
Other Adverse Events (participants affected / at risk) | 0/24 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT03980808/Prot_001.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT03980808/SAP_002.pdf
  • Informed Consent Form (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT03980808/ICF_003.pdf